CLINICAL TRIAL: NCT00227708
Title: Phase II Trial Assessing the Impact on Instrumental and Daily Living Autonomy of a Chemotherapy Regimen With Bi-Weekly Docetaxel in the Treatment of Metastatic or Locally Advanced Non-Small Cell Lung Cancer in Patients Over the Age of 70
Brief Title: Docetaxel in Treating Older Patients With Locally Advanced or Metastatic Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UNICANCER (Other)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000443593; FRE-FNCLCC-GERICO-05/0501; EU-20521
Record Dates: First submitted 2005-09-26; First posted 2005-09-28 (Estimated); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Lung Cancer
Keywords: adenocarcinoma of the lung; adenosquamous cell lung cancer; large cell lung cancer; squamous cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; recurrent non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Adenocarcinoma of Lung; Carcinoma, Non-Small-Cell Lung | interventions — Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: docetaxel
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as docetaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Chemotherapy drugs may have different effects in older patients.

PURPOSE: This phase II trial is studying how well docetaxel works in treating older patients with locally advanced or metastatic non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the quality of life of older patients with locally advanced or metastatic non-small cell lung cancer treated with docetaxel.

Secondary

* Determine the response rate in patients treated with this drug.
* Determine the overall survival and progression-free survival of patients treated with this drug.
* Determine the mood status and autonomy of activity of patients treated with this drug.
* Determine the toxicity of this drug in these patients.

OUTLINE: This is a multicenter study.

Patients receive docetaxel IV twice in week 1. Treatment repeats every 2 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed during study therapy in weeks 3-4, 7-8, and 11-12, and then at 6 and 12 months after completion of study treatment.

PROJECTED ACCRUAL: A total of 58 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed non-small cell lung cancer, including adenocarcinoma, squamous cell carcinoma, large cell carcinoma, or combination of these histologies

  * Stage IIIB (i.e., pleural T4) disease
  * Stage IV disease
  * Recurrent disease after prior surgery or radiotherapy allowed provided disease is in an area that was not previously irradiated
* Measurable disease by CT scan or MRI
* No symptomatic brain metastasis
* Activity of Daily Living Scale score ≥ 4
* Instrumental Autonomy of Daily Living Scale score ≥ 4

PATIENT CHARACTERISTICS:

Age

* 70 and over

Performance status

* Not specified

Life expectancy

* More than 3 months

Hematopoietic

* Neutrophil count > 1,500/mm^3
* Platelet count > 100,000/mm^3
* Hemoglobin > 10 g/dL

Hepatic

* Transaminases < 1.5 times normal
* Bilirubin normal
* Alkaline phosphatase < 2.5 times normal
* Pre-albumin > 1.5 mg/dL

Renal

* Creatinine clearance > 30 mL/min

Cardiovascular

* No congestive heart failure
* No unstable angina pectoris
* No myocardial infarction within the past year
* No uncontrolled hypertension
* No uncontrolled high-risk arrhythmias

Gastrointestinal

* No active peptic ulcer
* No inflammatory bowel disease

Neurologic

* No history of dementia or seizures that would preclude giving informed consent
* No peripheral neuropathy ≥ grade 2
* No history of significant neurologic disorders

Immunologic

* No history of hypersensitivity to the study drug or drugs formulated with polysorbate 80
* No active uncontrolled infection

Other

* No history of psychotic disorders
* No uncontrolled diabetes mellitus
* No absolute contraindication to corticosteroid use
* No other malignancy within the past 5 years except basal cell skin cancer or carcinoma in situ of the cervix
* No geriatric depression scale score ≥ 12/15
* No familial, social, geographical, or psychological reason that would preclude study follow up

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior chemotherapy for stage IIIB or IV non-small cell lung cancer
* No other concurrent chemotherapy

Endocrine therapy

* No concurrent chronic treatment with corticosteroids except low-dose (i.e., methylprednisolone ≤ 20 mg/day or equivalent) treatment that was initiated > 6 months ago

Radiotherapy

* See Disease Characteristics

Surgery

* See Disease Characteristics

Other

* More than 30 days since prior active participation in another therapeutic clinical trial
* No other concurrent anticancer therapy
* No other concurrent investigational drugs

Ages: 70 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2005-06; Study Completion 2006-08-29 (Actual)

PRIMARY OUTCOMES:
Quality of life

SECONDARY OUTCOMES:
Response rate
Overall survival
Progression-free survival
Mood status and autonomy of activity
Toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Fargeot, MD, Study Chair — Centre Georges Francois Leclerc
Locations (9):
- France (5):
  - Centre Medico-Chirurgical de Creil, Creil
  - Centre de Lutte Contre le Cancer Georges-Francois Leclerc, Dijon
  - Centre Hospitalier Intercommunal St. Aubin les Elbeuf, Elbeuf
  - Marseille Institute of Cancer - Institut J. Paoli and I. Calmettes, Marseille
  - Institut Curie Hopital, Paris
- Clinique De Genolier, Genolier, Switzerland
- United Kingdom (3):
  - Charing Cross Hospital, London, England
  - Centre for Cancer Research and Cell Biology at Belfast City Hospital, Belfast, Northern Ireland
  - West of Scotland Cancer Centre, Glasgow, Scotland